CLINICAL TRIAL: NCT03990116
Title: Efficacy of Lateral Kangaroo Care in Hemodynamic Stabilization of Premature Infant
Acronym: Cangulat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laura Collados Gomez (Other)
Responsible Party: Sponsor-Investigator, Laura Collados Gomez, Nurse at Neonatology Service, Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEO_nur_19
Record Dates: First submitted 2019-05-23; First posted 2019-06-18 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Kangaroo Care; Premature Infant; Body Temperature
Keywords: Patient Positioning; Kangaroo-Mother Care Method; skin to skin; Extremely Premature infant
MeSH Terms: conditions — Premature Birth | interventions — Prone Position

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lateral kangaroo (Experimental): Placing the infant in lateral on the parents chest, keeping the head neutral and limbs flexed towards body midline
  Interventions: Procedure: Lateral
- Prone Kangaroo (Active Comparator): placing the baby in upright and ventral position between mother's breasts or over the father chest, in skin-to skin contact with no clothes in between and with lower limbs flexed
  Interventions: Procedure: Prone

INTERVENTIONS:
Procedure: Lateral — Posture lateral kangaroo care
  Arms: Lateral kangaroo
Procedure: Prone — Posture prone kangaroo care
  Arms: Prone Kangaroo

SUMMARY:
The objetive of the study is to evaluate the non-inferiority or the equivalence of the kangaroo care position, in lateral versus traditional one in prone measuring the stability of several parameters in premature infants less than 28 weeks of gestational age during the first 5 days of life.

DETAILED DESCRIPTION:
A non-inferiority clinical trial, controlled, randomized and not blinded has been designed. The non-equivalent, experimental group consist on neonates less than 28 weeks of gestational age who are placed in lateral position while they are on kangaroo care during the first 5 days of life. On the other hand, the control group include neonates less than 28 weeks of gestational age who are in traditional prone position during kangaroo care on the first 5 days of life.

To define the sample size a power of 80% is assumed (β=0,20) and a 95% confidence interval (α=0,05) with a difference of 0,3ºC (SD 0,16) (9,10) in the axillary temperature. A non inferiority margin of 0.2ºC is established and a 10% sample size loss has been assumed. So a sample size of 35 premature in each group has been estimated.

A non probabilistic and consecutive sampling has been defined. The allocation into the experimental (lateral position) or control group (prone position) is going to be randomized.

The main outcome variable is the axillary temperature. However other clinical variables as pain, changes in the vital signs, HIV incidence rate are going to be measured as well.

ELIGIBILITY:
Inclusion Criteria:

* Premature under 28 weeks of gestational age with mother / father who wants kangaroo care.

Exclusion Criteria:

* Premature infants with mechanical ventilation in high frequency mode,
* Premature infants in the immediate postoperative period of major surgery,
* Premature infants with malformations of the abdominal Wall
* Premature infants who require immobilization
* Premature infants who do not tolerate kangaroo care: hemodynamic, thermal instability or increased stress
* Premature infants with duration of kangaroo care of less than 60 minutes.
* Also excluded are those patients where the kangaroo care provider has an anatomical limitation for carrying out kangaroo care.

Ages: 1 Minute to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Change from skin temperature | T0: baseline; T1: 30 minutes after to start kangaroo care; T2: 30 minutes after to finish kangaroo care
  Change from skin temperature after kangaroo care Peripheral temperature of the premature measured in the axilla with Braun® PRT2000 thermometer and the continuous temperature monitoring sensor of Giraffe ® incubators (AirLife TM infant skin temperature probe)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Collados, phD, Principal Investigator — Hospital Universitario 12 de Octubre
Locations (1):
- Laura Collados Gómez, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Collados-Gomez L, Esteban-Gonzalo L, Lopez-Lopez C, Jimenez-Fernandez L, Piris-Borregas S, Garcia-Garcia E, Fernandez-Gonzalo JC, Martinez-Miguel E. Lateral Kangaroo Care in Hemodynamic Stability of Extremely Preterm Infants: Protocol Study for a Non-Inferiority Randomized Controlled Trial CANGULAT. Int J Environ Res Public Health. 2021 Dec 28;19(1):293. doi: 10.3390/ijerph19010293. PMID 35010554